CLINICAL TRIAL: NCT02568774
Title: Acupuncture on Post-Stroke Overactive Bladder: A Randomized Controlled Trial
Brief Title: Acupuncture on Post-Stroke Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Haiyong Chen, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AcupPSOAB
Record Dates: First submitted 2015-06-13; First posted 2015-10-06 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Overactive Bladder
Keywords: Post-stroke
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional Acupuncture (Experimental): Acupoints which are empirical for treating OAB in terms of Traditional Chinese medicine theory are used (in the sequence of scalp reproduction area and motor area of the unaffected side, RN3, bilateral BL32, BL33, BL28, BL39). And Ear point urinary bladder, and Ear point uterus will be treated after removal of needles. Needles will be left for 30 minutes and then removed. Subjects will be treated with acupuncture 2 times per week for the first 2 weeks and 1 per week for the 3rd and 4th week.
  Interventions: Other: Traditional Acupuncture
- Usual Care (Other): Patients will receive conventional rehabilitation as usual, including standard physiotherapy, bladder training and general advise of fluid intake.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Traditional Acupuncture — Treatment is based on the traditional Chinese medicine theory for treating overactive bladder. Qi-transforming function of bladder is regulated by experienced Chinese medicine practitioner.
  Arms: Traditional Acupuncture
Other: Usual Care — Patients will receive conventional rehabilitation as usual, including standard physiotherapy, bladder training and general advise of fluid intake.
  Arms: Usual Care

SUMMARY:
This study evaluates the effect of acupuncture on post-stroke overactive bladder symptoms. Participants will be put into groups randomly and compared. There are two groups: traditional acupuncture and usual care. The ratio of group allocation is 1:1.

DETAILED DESCRIPTION:
Current practice in management of OAB is quite limited. Acupuncture, which is a major treatment modality of traditional Chinese medicine, has also claimed to have favourable therapeutic effect on OAB. Previous study found that acupuncture at the BL-33 point was effective for controlling the overactive bladder. Although acupuncture has been shown to be effective in treating OAB, there has been no randomized controlled trial examining the efficacy of acupuncture on patients with post-stroke. Given the high incidence of OAB in post-stroke patients, potentially effective alternative treatments should be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese aged 18 or above
2. Patient suffering from first ever stroke or recurrent stroke with no urinary symptom in previous episode(s);
3. Patient with classic symptoms, i.e. urgency, urinary frequency or urge incontinence and Overactive Bladder Symptom Score (OABSS) score ≥3 and the urgency item rated as at least 2-point;
4. Not taking any medication for OAB
5. Able to communicate
6. No current acupuncture or transcutaneous electrical nerve stimulation treatment

Exclusion Criteria:

1. Urinary retention with post-void urinary volume > 100ml;
2. Current urinary tract infection;
3. Preexisting history of OAB or bladder outlet obstruction or underactive bladder;
4. Significant cognitive impairment with MMSE < or =19;
5. Coexisting Alzheimer's disease, Parkinson's disease, spinal cord disorder or progressive neurological disease such as multiple sclerosis;
6. Active skin lesion or open wound over the needle placement areas;
7. Having valvular heart defects, severe cardiac diseases, or bleeding disorders,
8. Being fitted with any implanted electrical device such as pacemaker, defibrillator, or brain stimulation;
9. Pregnant;
10. Malignancies at the sites of selected acupoints;
11. Receiving acupuncture treatment 1 month before baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-08; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Overactive Bladder Symptom Scale (OABSS) | 1-week posttreatment
  four item questionnaire quantifies overactive bladder symptoms in a single score

SECONDARY OUTCOMES:
Number of incontinent episodes measured by bladder diary | 1-week posttreatment, 4-week posttreatment
  Record the frequency of day and night time voiding and incontinence episodes over 3 day periods
Stroke Specific Quality of Life Scale (SS-QoLS) | 1-week posttreatment, 4-week posttreatment
  12 items questionnaire consists of physical and psychosocial subscales: amount of help required completing a task, trouble experienced performing a task and functioning.
Medication measured by bladder diary | 1-week posttreatment, 4-week posttreatment
  number of patients requested medication for OAB from bladder diary.

OTHER OUTCOMES:
AE measured by open-ended questions | first week of treatment, second week of treatment, third week of treatment, 1-week posttreatment, 4-week posttreatment
  open-ended questions about the experience of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Wing Fai Yeung, BCM, PhD, Principal Investigator — The University of Hong Kong
Locations (3):
- Shanghai TCM-INTEGRATED Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai, China
- Hong Kong (2):
  - Tung Wah Eastern Hospital, Hong Kong
  - Tung Wah Hospital, Hong Kong